CLINICAL TRIAL: NCT00265720
Title: Research on Community Cancer Control: Study of Colorectal Cancer Screening in the African American Population
Brief Title: Colorectal Cancer Screening Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator: D. Blumenthal, Morehouse School of Medicine
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: H57/CCH420680-05; H57/CCH420680-05
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer; Colorectal Cancer Screening
Keywords: African Americans; Colorectal Cancer Screening; Colorectal Cancer; Colorectal Cancer and African Americans; Cancer Disparities
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Written materials only
  Interventions: Other: Control
- Reduced out-of-pocket expense (Experimental): Reimbursed up to $500 out-of-pocket expense for colorectal cancer screening
  Interventions: Other: Reduced out of pocket expense
- One-on-one education (Experimental): Individual education with a health educator on CRC screening
  Interventions: Behavioral: one on one education
- Group Education (Experimental): Education on CRC screening in a small group with a health educator
  Interventions: Behavioral: Group education

INTERVENTIONS:
Other: Control — Written materials only
  Arms: Control
Other: Reduced out of pocket expense — Reimbursed up to $500 out of pocket expense for CRC screening
  Arms: Reduced out-of-pocket expense
Behavioral: one on one education — one on one education with a health educator
  Arms: One-on-one education
Behavioral: Group education — Education in a small group
  Arms: Group Education

SUMMARY:
Colorectal cancer is the second deadliest among cancers and disproportionately affects African Americans. The Colorectal Cancer Screening Intervention Trial(CCSIT) project has as its goal to test three interventions designed to increase screening rates among medically underserved African Americans in the Metropolitan Atlanta area. It is designed to increase awareness of modifiable risk factors and promote the benefits of screening as a means of early detection of colorectal cancer. mportance of being screened for colorectal cancer,African Americans continue to be disproportionately affected by this disease. The Colorectal Cancer Screening

DETAILED DESCRIPTION:
Despite increased awareness of the importance of being screened for colorectal cancer, African Americans continue to be disproportionately affected by this disease. The Colorectal Cancer Screening Intervention Trial (CCSIT) is designed to test and expand a public health intervention that combines social marketing and community-coalition building efforts.

The purpose of this study is to 1) evaluate the effects of three different approaches on knowledge, attitudes and beliefs (KABs) about colorectal cancer; 2) to examine the effects of three different approaches to adherence to screening guidelines and 3) to evaluate the independent role of setting on screening practices.

Participants age 50 and over are recruited from churches, clinics and senior sites which allows us to examine the impact of setting on participant recruitment and changes to KAB. Pre and post questionnaires are administered to determine the knowledge attitudes and behaviors (KAB) related to screening and to measure psychosocial parameters (self-esteem, perceived stress and social support). These persons are randomized into one of four groups, the control group and three intervention arms: (1) one-on-one counseling sessions, (2) small group educational sessions and (3) financial incentives interventions where out of pocket cost for screening is reimbursed. The counseling and educational interventions incorporate the Health Belief Model and Social Learning Theory.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Previously not screened for colorectal cancer according to ACS guidelines
* Reside in Fulton,,Gwinett,Cobb,Clayton and DeKalb counties
* 50 years of age or older

Exclusion Criteria:

* Non-African American
* Less than 50 years of age
* Previously screened consistent with ACS guideline

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening Rate; This measurement(Impact) is taken 90 days from last intervention session. If a person is not screened, an additional measurement(Post-Impact) is taken 90 days from the Impact.

SECONDARY OUTCOMES:
Knowledge, Attitudes and Beliefs; this measurement is taken at baseline and post intervention session. Sessions vary by intervention group after the initial recruitment sessions:

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumenthal, M.D., M.P.H., Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- See also: Morehouse School of Medicine - Prevention Research Center — http://www.msm.edu/prc/